CLINICAL TRIAL: NCT01021098
Title: A Multi-center Military Consortium for Clinical Research Into the Natural History, Host Response, and Potential Therapy of Acute Respiratory Infection in Military Members and Their Families
Brief Title: Acute Respiratory Infection Consortium
Acronym: ARIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IDCRP-045; HT9404-12-2-0004 (Other: National Institute of Allergy and Infectious Diseases)
Record Dates: First submitted 2009-11-10; First posted 2009-11-26 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Influenza
Keywords: influenza; illness; active-duty; virus; flu; military; Influenza-like-illnesses
MeSH Terms: conditions — Influenza, Human; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — nasal swabs with storage of multiple harvested (expanded) first generation viral isolates (all must opt in); buccal swab storage (may opt out) rectal swab storage (may opt out) serum storage (may opt out)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Natural History Study: The core Natural History Study of ILI is an observational, longitudinal cohort study using data from clinical findings, medical chart review, and diagnostic, virologic and immunologic laboratories to describe the epidemiology and immunology of ILI. This study aims to describe the clinical history of influenza and other viral respiratory pathogens in a population of US military active duty members and their dependents. The primary focus will be the etiology, natural history and immunology of ILI in otherwise healthy adults and children. We will recruit subjects with ILI in both the outpatient and inpatient setting, and will serially collect biological specimens (e.g. nasal/throat swabs, blood, rectal swabs) over a 28-day period. In addition, we will collect a single buccal (cheek) swab.
- HIV-Positive Cohort: In addition, given a number of human immunodeficiency virus (HIV)-infected subjects who serve in the active duty force, we will also examine a subset of HIV-positive military beneficiaries as part of this consortium. An additional objective of the study will be to descriptively examine the clinical and laboratory characteristics of ILI events among HIV-infected persons using the military's substantial experience in following a stable HIV-infected population. We will recruit subjects with ILI in both the outpatient and inpatient setting, and will serially collect biological specimens (e.g. nasal/throat swabs, blood, rectal swabs) over a 28-day period. In addition, we will collect a single buccal (cheek) swab.

SUMMARY:
Recently, the emergence and rapid global dissemination of novel swine-origin influenza A virus (H1N1) with unique epidemiologic characteristics has heightened awareness and concern of this viral pathogen, and its potential for major disruption of both civil and military stability. Although advances in medical and scientific technologies have improved our basic understanding of respiratory disease, many questions about the epidemiology and immunology of ARI remain unanswered. This study plans to initiate a multi-site, multi-disciplinary research collaboration, termed the Acute Respiratory Infection Consortium (ARIC) for the purpose of studying the etiology, epidemiology and immunology of influenza-like illness (ILI) in order to describe the natural history and risk factors for disease, as well as the characteristics of the host immune response.

At the core of the ARIC is the proposed observational, longitudinal study of the Natural History Study of ILI among active duty military members, healthy retirees, and their dependents recruited from both inpatient and outpatient settings of military treatment facilities (MTF) in the continental US to be followed for a total of four (4) visits over a 28-day period. Additionally, the investigators also propose to conduct a household-based study of influenza (Family Transmission Study) in which individuals who have a laboratory-confirmed influenza illness will be recruited and enrolled along with their family members for the purpose of studying transmission of influenza within households. Taken together, these studies will establish a longitudinal cohort of ILI among active duty members and their families, as well as a repository of biological specimens relevant to the epidemiology and immunology of infection. Ultimately, these studies will serve as a solid foundation on which future investigations of ARI epidemiology, treatment and prevention can be based.

DETAILED DESCRIPTION:
This is an observational, longitudinal study of ARI/ILI among otherwise healthy active duty military members, retirees, as well as their spouses and dependents. An additional cohort of HIV-infected adults will also be evaluated. We will collect data from clinical findings, medical chart review, and diagnostic, virologic, and immunologic assays to describe the epidemiology and immunology of ARI/ILI. Subject recruitment will take place in both inpatient and outpatient settings of military treatment facilities (MTF) in the continental US. Additionally, subject self-referral will be encouraged through institutional review board (IRB) approved advertisements. Both adults under 65 years of age and children will be eligible for participation. Subjects will be followed for a total of up to 4 visits over a 28±7-day period. After their final visit (Day 28±7 applicable window), participants may only re-enroll into the study after 3 months have passed.

Nasal swabs, blood specimens (if consented to), buccal cytobrush samples (if consented to), and rectal swabs (in select subgroups of consenting inpatients) will be collected in order to characterize the etiologic, epidemiologic, and immunologic characteristics of ARI in the study population. In the HIV- positive cohort, additional clinical data and blood will be collected for HIV-specific factors (e.g., CD4 counts, HIV RNA levels) and for additional immunologic studies at days 0 and 28 (± 7) of the study. This is a prospective longitudinal study which will use data from clinical findings, medical chart review, and diagnostic, virologic and immunologic laboratories to describe the epidemiology and immunology of ARI/ILI.

ELIGIBILITY:
Natural History Study

Inclusion Criteria:

* Between 18 and 55 years of age (inclusive), or a 17 year old military service member
* Eligible for care in Department of Defense (DOD) facilities (DEERS eligible).
* Have an acute influenza-like illness (ILI) or severe acute respiratory infection (SARI) for </= 7 days

Exclusion Criteria:

* None

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Males and females ages 17-55 and of military (including active duty enlisted and active duty officers from all branches of service), healthy retirees, and their dependents (spouses and children) presenting to inpatient/outpatient facilities with ILI will be eligible for participation. 17 year old enrollees must be active duty and therefore considered adults per DoDI 3216.02.
Sampling Method: Probability Sample
Enrollment: 2018 (Actual)
Dates: Start 2009-11; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of subjects enrolled in the IDCRP ARI Consortium Natural History Study | 10 years
  Clinical signs and symptoms,antibody titers (sera), serum cytokines and cell-mediated immunity (peripheral blood mononuclear cell activity), along with pathogen data (nasal swab/fecal swab), human leukocyte antigen (HLA) using a buccal swab, and fecal swabs to study the epidemiology, etiology , clinical characteristics and immunology of medically-attended ILI and SARI cases in this population.

SECONDARY OUTCOMES:
Develop and validate a patient-reported influenza outcome (Flu-PRO) instrument in patients with influenza-like illness | 6 months
  Internal consistency reliability of the Flu-PRO Total and Domain scores on day 1
Impact of HIV-status on symptom severity, as measured by mean total composite score using Flu-Pro instrument, in subjects with influenza-like-illness | 1 year
  Mean total composite symptom scores during the ILI episode were compared by HIV status using multivariate linear models, controlling for other factors such as influenza season, age, race, and military status. Measurement tool = Flu-Pro
Describe patterns of viral shedding by viral pathogen and pathogen subtype | 1 year
  Serial nasal swabs collected from patients will be used to determine the duration of viral shedding

CONTACTS AND LOCATIONS:
Overall Officials: Timothy H Burgess, MD, MPH, Principal Investigator — Uniformed Services University of the Health Sciences/Infectious Disease Clinical Research Program
Locations (5):
- United States (5):
  - Naval Medical Center, San Diego, CA, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - San Antonio Military Medical Center/Wilford Hall, San Antonio, Texas
  - Naval Medical Center, Portsmouth, VA, Portsmouth, Virginia
  - Madigan Army Medical Center (MAMC), Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
We plan to directly share de-identified data with the third party Menssana Research Inc. for a substudy of an investigational device for the diagnosis of influenza. This data will include basic demographic information, flu diagnostic results, smoking status, and symptom history. This data will be de-identified and shared directly with the third party via secure file transfer. This applies only to participants recruited into the substudy at the site San Antonio Military Medical Center.
Time Frame: 2018 to 2020
Access Criteria: Researchers are required to submit a formal request describing the research questions of interest and protocol for review. If the request is approved, IDCRP investigators must be listed on any research publications resulting from research using the study data.

REFERENCES:
- [Derived] Colombo RE, Schofield C, Richard SA, Fairchok M, Chen WJ, Danaher PJ, Lalani TN, Ridore M, Maves RC, Arnold JC, Ganesan A, Agan B, Millar EV, Coles C, Burgess TH. Effects of human immunodeficiency virus status on symptom severity in influenza-like illness in an otherwise healthy adult outpatient cohort. J Investig Med. 2021 Aug;69(6):1230-1237. doi: 10.1136/jim-2020-001694. Epub 2021 Apr 23. PMID 33893210
- [Derived] Deiss RG, Arnold JC, Chen WJ, Echols S, Fairchok MP, Schofield C, Danaher PJ, McDonough E, Ridore M, Mor D, Burgess TH, Millar EV. Vaccine-associated reduction in symptom severity among patients with influenza A/H3N2 disease. Vaccine. 2015 Dec 16;33(51):7160-7167. doi: 10.1016/j.vaccine.2015.11.004. Epub 2015 Nov 10. PMID 26562321